CLINICAL TRIAL: NCT01304745
Title: Rehabilitation of Women Following Treatment for Gynaecological Cancer; a Randomized, Controlled Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2009/896
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Gynecologic Cancer
MeSH Terms: interventions — Population Groups; Exercise; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Physical traning in group (Experimental)
  Interventions: Behavioral: Physical training in group
- Educational and counselling group (Experimental)
  Interventions: Behavioral: Educational and counseling in group
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Physical training in group — Physical training in group, 6-9 participants, two times av week (1.5 hours) over a period of 16 weeks, focusing on strength and endurance training including body awareness and relaxation.
  Other Names: Physical exercise
  Arms: Physical traning in group
Behavioral: Educational and counseling in group — Educational and counseling groups with 6-9 participants, with seven group meetings 2.5 hours over a period of seven weeks. Each session starts with a (20 minutes) lecture were one out of seven different topics are presented (Fatigue, sexuality, coping and coping strategies, etc).
  Other Names: nurse-led patient education
  Arms: Educational and counselling group

SUMMARY:
The purpose of the study is to evaluate and compare the effect of: 1 Educational and counselling in groups, 2) Physical training in group with 3) Control group, on global- and health related quality of life and coping in patients finished treatment for gynaecological cancer.

DETAILED DESCRIPTION:
Previous studies have shown that gynaecological cancer patients may suffer from both psychological and physiological long term side-effects. Cancer surgery, radiotherapy and chemotherapy may result in physical symptoms like gastro-intestinal problems and related pelvic pain (White, 2008).

The persons quality of life may also be influenced after finished cancer treatment and may be manifested with both physical and psychological problems such as fatigue (subjective experience of fatigue and lack of energy) (Vistad et al., 2007), anxiety and depression, sleep problems and fear of relapse (Lagana et al., 2001, Wenzel et al., 2002, Hodginson, 2007). The concept of quality of life is something different operationalized and defined across different studies. In the present study the quality of life will be defined from both global- and health related quality of life. The physical and psychological after-effects of the treatment also influences the social function, and hence the ability to get back to work (Boer et al., 2009). It generally agreed that a high proportion of women of working age do not come back to work after undergone cancer treatment. The women's experience of returning to work, according to Kennedy et al. (2007), is a unknown area of cancer research.

Previous research have shown that participation in educational-, counselling- and physical training groups may have positive effects on the quality of life for women treated for gynaecological cancer. As far as we know, however, no randomized controlled studies have measured and compared the effects of both educational and counselling intervention versus physical training in groups on women's self-reported quality of life and coping. The purpose of this study is therefore to evaluate and compare the effect of educational- and counselling in groups and physical training in groups on women's self reported quality of life and coping.

The present study is a collaboration between Haukeland University Hospital (HUH), Bergen University College, University of Agder, University of Stavanger, Stavanger University Hospital and Sørlandet Hospital. The study is carried out between 2009 and 2013. The participants diagnosed and treated for gynaecological cancer between January 2007 - January 2012 received/will receive a information letter and informed consent per post or during the regular follow-up appointments at the Hospitals. All women fulfilling the inclusion criteria and finished treatment at HUH between January 2007 and to January 2012 are invited/will be invited to participate in the present study. At Stavanger University Hospital and Sørlandet Hospital patients finished treatment form 2008 is invited to participate in the present study.

This intervention study has a randomized controlled design with: 1) Educational and counselling groups, 2) Physical training in a group, 3) Control group, with three repeated measures at pre- intervention, post-intervention and at 1-year follow-up. The educational and counselling groups have one session a week over a period of seven weeks. The physical training groups have two sessions a week for 16 weeks, focusing on strength and endurance training. The control group follows only the standard post-treatment procedure at the specific Hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Women finished treatment with a curative purpose independent of stage of cancer, type of gynaecological cancer, or previous gynaecological cancer
* Meet a certain physical functioning criteria (Specified as; manage to walk 3.1 miles per hour, lie down and rise up from the floor)
* To be willing to participate in the study for a period of 1- year and agrees to participate as specified conditions according to the consent form
* Not having any significant amnesic symptoms
* Women with other diagnosis were included as far as criterion 3 was fulfilled

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2009-10; Primary Completion 2013-09 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Global- and health related quality of life | Pre intervention, post intervention and at one year follow-up

SECONDARY OUTCOMES:
Coping strategies after gynaecological cancer | Pre intervention, post intervention and at one year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Margrethe Vika, AP, Principal Investigator — Haukeland University Hospital
Locations (1):
- Margrethe Vika, Bergen, Norway